CLINICAL TRIAL: NCT06599034
Title: Strategies to Increase Adherence to Physical Activity in a Phase III Cardiac Rehabilitation Program
Status: Completed | Type: Observational
Sponsor: Hospital de Manises (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-132-1
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ischaemic Heart Diseases
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study consists of a randomised clinical trial of two parallel groups conducted in patients with ischaemic heart disease after completing phase II of Cardiac Rehabilitation (RHBC) at the Centro de Especialidades Mislata (CEM),Hospital Manises. The objective is to assess adherence to structured and unstructured physical activity in the long term (6 and 12 months). In addition to the usual recommendations in the Control Group (CG), a motivational programme will be added to the Intervention Group (IG), which will consist of establishing an individualised exercise plan reviewed monthly, in addition to maintaining continuous contact with the physiotherapist.

DETAILED DESCRIPTION:
Regular physical activity is an important measure in the prevention of cardiovascular diseases. In the phase II Cardiac Rehabilitation programme, the acquisition of healthy lifestyle habits is taught and encouraged, with physical exercise as a fundamental pillar of the programme. Physical exercise should be maintained throughout life (RHBC phase III) in order to continue to produce cardiovascular benefits. However, few studies focus on strategies to increase adherence to physical activity, despite its benefits in disease control.

Motivation is one of the main barriers described by patients as well as the lack of contact with healthcare staff once the acute disease process is over. Therefore, we propose a simple, practical and economical intervention to increase adherence to physical activity, through a motivational programme, based on the establishment of objectives for each patient, carrying out an individualised physical exercise programme according to their preferences and needs, also establishing continuous contact with the physiotherapist to review and establish new objectives.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischaemic heart disease who have completed phase II of cardiac rehabilitation in CEM.
* Patients of both sexes.
* Patients classified as low, medium and high risk
* Age between 18 and 70 years at the time of the cardiac event.

Exclusion Criteria:

* Older 70 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is all patients with ischaemic heart disease who have completed phase II in the Cardiac Rehabilitation Service of Centro de Especialidades Mislata, Hospital Manises.
  The final sample is made up of patients who have completed all the sessions of the cardiac rehabilitation programme (20 sessions for high-moderate risk patients, 16 sessions for low-risk patients) and meet all the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Patient Adherence to Physical Activity | The groups, CG ad IG, will be assessed at four times: at baseline, at finish of the phase II CRP, at 6 months after the finish phase II CRP and at 12 months after the finish of phase II CRP.
  Registry of the characteristics of physical exercise following the principle: frequency, intensity, time and type of exercise
Participants Adherence to Physical Activity. Steps Control | The groups, control group (CG) and intervention group (IG), will be assessed at two times, 6 months and 12 months after the finish phase II of cardiac rehabilitation program (CRP).
  Registry of daily physical activity, steps per day, by means of an OMROM HJ-321-E pedometer

SECONDARY OUTCOMES:
Changes in Functional Capacity: measurement of ergometer | The groups, CG and IG, will be assessed at three times: at baseline, at finish phase II cardiac rehabilitation program, at 12 months after the finish phase II CRP.
  Incremental of ramp protocol exercise text in a treadmill
Changes in Blood Pressure | The groups, CG and IG, will be assessed at four times: at baseline, at finish of the phase II CRP, at 6 months after the finish phase II CRP and at 12 months after the finish of phase II CRP
  Blood pressure recording using an OMROM HcM-FC 31 blood pressure monitor
Changes in biochemical variables | The groups, CG and IG, will be assessed at three times: at baseline, at finish phase II cardiac rehabilitation program, at 12 months after the finish phase II CRP.
  Registry of the values of total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, basal glycaemia and glycosylated haemoglobin to be analysed by means of a blood test
Changes in abdominal circumference | The groups, CG and IG, will be assessed at four times: at baseline, at finish of the phase II CRP, at 6 months after the finish phase II CRP and at 12 months after the finish of phase II CRP.
  Registry of centimetres of abdominal circumferene, midpoint from the lower rib margin to the antero-superior iliac crest in standing position, using measuring tape.
Changes in Muscle Mass Index( BMI) | The groups, CG and IG, will be assessed at four times: at baseline, at finish of the phase II CRP, at 6 months after the finish phase II CRP and at 12 months after the finish of phase II CRP.
  Weight (kg) and height (m) will be recorded
Changes in the perception of quality of life | The groups, CG and IG, will be assessed at four times: at baseline, at finish of the phase II CRP, at 6 months after the finish phase II CRP and at 12 months after the finish of phase II CRP
  Registry of the score obtained by means of the SF-12 quality of life questionnaire, in its version adapted and validated in Spanish
Changes in anxiety levels | The groups, CG and IG, will be assessed at four times: at baseline, at finish of the phase II CRP, at 6 months after the finish phase II CRP and at 12 months after the finish of phase II CRP.
  Registry of the score obtained from the State-Trait Anxiety Questionnaire (STAI) in its version adapted and validated in Spanish
Changes in depresión levels | The groups, CG and IG, will be assessed at four times: at baseline, at finish of the phase II CRP, at 6 months after the finish phase II CRP and at 12 months after the finish of phase II CRP
  Registry of the score obtained in the Beck Depression Inventory-II (BDI-II) in its version adapted and validated in Spanish

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Manises, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No